CLINICAL TRIAL: NCT04391998
Title: Parasitic Infection in Anemic Pregnant Women. Prevalence and Effects in Rural Area in Egypt.
Brief Title: Parasitic Infection in Anemic Pregnant Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, PROFESSOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 175
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Anemia of Pregnancy
MeSH Terms: interventions — Iron-Dextran Complex; Metronidazole; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anemia without parasitic infection (Active Comparator): women with anemia without parasitic infection will receive iron treatment
  Interventions: Drug: Iron Supplement
- parasitic infection treated with iron (Active Comparator): women with anemia with parasitic infection will receive oral iron treatment
  Interventions: Drug: Iron Supplement
- parasitic infection treated with iron and antihelmemsic (Active Comparator): women with anemia with parasitic infection will receive oral iron treatment and antihelminsic treatment in the form of metronidazole 500mg tab twice daily for 5 days in cases with Entamoeba or Giardia or albendazol 200mg tab
  Interventions: Drug: Iron Supplement; Drug: Metronidazole Oral; Drug: Albendazole

INTERVENTIONS:
Drug: Iron Supplement — oral tablet twice daily after meals
  Other Names: Ferroglobin
Drug: Metronidazole Oral — 500 mg oral twice daily
  Other Names: Flagyl
  Arms: parasitic infection treated with iron and antihelmemsic
Drug: Albendazole — 200 mg oral single dose
  Other Names: alzental
  Arms: parasitic infection treated with iron and antihelmemsic

SUMMARY:
Women included between 18 and 45 years old, pregnant during their second or third trimester of pregnancy (calculated by a sure menstrual date and confirmed by a 1st trimesteric ultrasound) with hemoglobin level below 10.5 mg /dL.

DETAILED DESCRIPTION:
All patients in the study were subjected to:

1. Detailed history was recorded. A proper history concerning age, sex, residence, socioeconomic status, onset, progression, and previous treatment of anemia was taken. Participants' socio-demographic characteristics including gravida and parity were documented, level of education, occupation, Diet, and information useful to determine the socioeconomic level was recorded. Information on previous pregnancies and children and history of chronic diseases were also recorded.
2. General examination; patients were clinically examined and gestational age (assessed by measuring the fundal height), weight was calculated for each participant.
3. Diagnosis of anemia by Complete blood count (CBC), Hb level and measuring hematocrit concentration.
4. Diagnosis of parasitic infection by stool analysis using suitable techniques.
5. Imaging including obstetric ultrasound (U/S) to assess fetal development.
6. Women with helminthic infections will be divided into groups

Group (A): received iron + antiparasitic treatment as follows:

* Patients who have STH received alzental 200mg tab 2 tabs single oral dose.
* Patients who have Entamoeba or Giardia received flagyl 500mg tab twice daily for 5 days.
* (B): received iron only.

ELIGIBILITY:
Inclusion Criteria:

* pregnant during their second or third trimester of pregnancy (calculated by a sure menstrual date and confirmed by a 1st trimesteric ultrasound)
* hemoglobin level below 10.5 mg /dL

Exclusion Criteria:

* women with chronic diseases as diabetes, heart, renal, hepatic or endocrinological disorders
* women diagnosed with blood diseases as hemoglobinopathy or vascular diseases as vasculitis.
* Women with autoimmune diseases and those allergic to iron or antihelminsic treatment were also excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
correction of naemia | 6 weeks after treatment
  hemoglobin level increased above 11 gm/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided